CLINICAL TRIAL: NCT05852483
Title: Perioperative Predictors of Postoperative Readmission Among Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Predictors of Readmission in Patients Undergoing PNL
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hazem Tarraf Abo Dief, principal investigator, Assiut University
Other Study IDs: Post PNL readmission
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2023-05

CONDITIONS: Kidney Stone
Keywords: Predictors, Percutaneous nephrolithotomy, Readmission
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To identify predictors of patients postoperative readmission after PNL

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is a minimally-invasive procedure to remove stones from the kidney by a small puncture wound (up to about 1 cm) through the skin. It is usually done under general anesthesia or spinal anesthesia. Despite the advancements in endoscopic technologies technique and training, the procedure is still associated with complications, which can occur during the intervention or in the early or late postoperative period. Known complications to PCNL are fever (2.8-32.1%), bleeding requiring transfusion (0- 45%), organ injury (0-1.7%) and sepsis (0.3-1.5%) these complications consider life threatening and increase risk of patient readmission Readmission is defined as a state when the patient is admitted to the same or a different hospital after being discharged from the applicable hospital to a non-acute setting, such as his home within a specified time period . Hospital readmissions are frequent and costly, and are estimated to cost the US health care system > $12-17 billion annually . Readmissions occurring within the first week after discharge are often related to the stress of acute illness as well as heightened self-care needs, new medications, and impaired function while those occurring later reflect chronic illness Nurses could play a pivotal role in preventing readmissions through appropriate discharge teaching and following up with the patients after discharge through telephone conversations. Early identification of patients' problems and taking appropriate measures to handle these problems at an early stage helps to prevent further post-discharge complications and improves patient outcomes.

Nurse should emphasize to the patient the importance of reporting symptoms to physician immediately. Postoperative care should include: close monitoring of vital signs, close observation of urine output and color changes, wound care and careful observation for dressing and tube drainage.

Many studies have been found in the literature on readmissions after urological surgeries and their causes in recent years . These studies include general urological surgical procedures, and there are limited studies examining potential predictive factors for endourology and stone surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients
* patients shechedled for PNL
* age range from)18-65(years

Exclusion Criteria:

* Failed PNL
* psychiatric patients
* coagulopathy
* patients refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult male and female patients who had undergone PNL and their age range from)18-65(years in Assiut governorate
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
comparison between readmitted and non readmitted regarding readmission risk factors | baseline
  analysis preioperative factors that lead to readmission after PNL

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of nursing, Assiut University, Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma K, Sankhwar SN, Goel A, Singh V, Sharma P, Garg Y. Factors predicting infectious complications following percutaneous nephrolithotomy. Urol Ann. 2016 Oct-Dec;8(4):434-438. doi: 10.4103/0974-7796.192105. PMID 28057987
- See also: Members of the European Association of Urology (EAU) Guidelines Office. Guidelines on urolithiasis. 2019 — http://uroweb.org/guideline/urolithiasis